CLINICAL TRIAL: NCT01318785
Title: Therapeutical Assessment of Compression Armsleeves for Lymphatic Indications (Therapeutische Bewertung Von Armkompressionsstrümpfen für Lymphatische Indikationen BF09-PH-01)
Brief Title: Therapeutical Assessment of Compression Armsleeves for Lymphatic Indications
Acronym: BF09-PH-01
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medicine Greifswald (Other)
Collaborators: KABEG Management (Other); Nij Smellinghe Hosptial (Other); Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Prof. Dr. med. Michael Jünger, Klinik und Poliklinik für Hautkrankheiten der Universität Greifswald
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Multicentrestudy "BF09-PH-01"
Record Dates: First submitted 2010-12-03; First posted 2011-03-18 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Lymphedema
Keywords: secondary arm-lymphedema; breast cancer related arm-lymphedema
MeSH Terms: conditions — Lymphedema; Breast Cancer Lymphedema

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Compression ArmsleevesType A (Active Comparator): Product A: armsleeves of type SoraLife KKl. 2 according to RAL GZ 387
  Interventions: Other: Compression Armsleeves
- Compression Armsleeves Type B (Active Comparator): Product B: armsleeves of type Elvarex KKl. 2 according to RAL GZ 387
  Interventions: Other: Compression Armsleeves

INTERVENTIONS:
Other: Compression Armsleeves — Type: Compression Class II (according to RAL)
  The study is designed in a way, that per product after a one weak resting (preparing) cycle a 2 weeks wearing period will follow. Herewith the whole duration of the study is 6 weeks per patient.
  Other Names: Bauerfeind SoraLife; Jobst Elvarex

SUMMARY:
Examination of therapeutical effects of different types of armsleeves in treating lymphatic diseases after breast cancer surgery during maintenance phase

1. thesis:

   - all types should be equal regarding volume reduction
2. thesis: armsleeves manufactured with microfibre yarn are expected to be

   * better in wearing comfort and
   * better in handling features.

DETAILED DESCRIPTION:
1. thesis:

   * measuring of arm volume by "inverse water-volumetry" (see later)
   * measuring of circumference cD
   * measuring of circumference cG
   * photodocumentation in 2 positions(during each round)
2. thesis

   * questionaire for patients

     * in the beginning
     * after 1 week
     * after 2 weeks (at the end of a wearing period)
   * questionaire for study nurse (at the end of a wearing period)

ELIGIBILITY:
Inclusion Criteria:

* women with a secondary arm-lymphedema for at least 3 months
* willingness to wear compression arm-sleeves for at least 12 hours per day
* maintenance phase, where no significant further reduction of arm-volume can be achieved
* lymphedema in stadium 1 or 2
* age: at least 18 years
* signed consent form by the patient
* sufficient knowledge in national language

Exclusion Criteria:

* edema not completely reduced to "maintenance phase"
* immobilized patient
* acute deep vein thrombosis in arm
* directly after arm-vein-thrombosis
* acute arm erysipelas
* malignant edema
* existent lipedema
* arterial occlusion
* distinctive neuropathy in upper limbs
* neurinoma in upper limbs
* chronic pain after plastic surgery in upper limbs, shoulder or breast
* change in drug treatment, that can influence edema situation during the study
* pregnant women
* breast giving mothers
* not signed consent form
* participation in a second clinical trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-09; Primary Completion 2011-10 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
change of volume (arm and hand together) | 6 weaks per patient
  During a 2-weeks-phase the volume of patients arm and hand together is measured once a week, e.g. 3 times (beginning, after 1 week, at the end).
  This is done with armsleeves of the first type. After one week of sedation the test will be repeated with the second product.
  Randomization is given by chance, that during first phase product of type A or type B can be applied. During second phase then vice versa.
  The measurements were performed by an "inverse water plethysmography device" (later: inverse watervolumetry) desinged by R. Damstra.

SECONDARY OUTCOMES:
Clinical judgement of skin status | 6 weaks per patient
  clinical judgement of skin status with photo documentation, clinical finding (as palpation,check on fibrosclerosis, skin clour, skin surface, edema, tenderness, tissue consistency...), check of skin contamination
Wearing comfort and handling features of armsleeves | 6 weeks per patient
  For both types of products questionaires are prepared to find out how patients are feeling with their armsleeves.It is asked for problems during donning procedure as well as during wearing period. This will be done in the beginning after 1 week and after 2 weeks for both types.
  At the end the study nurses are asked to their impression regarding patients acceptance of the armsleeves.
  Method: VAS score

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jünger, Prof. Dr., Principal Investigator — Klinik und Poliklinik für Hautkrankheiten der Universität Greifswald
Locations (4):
- Landeskrankenhaus Wolfsberg, Wolfsberg, Carinthia, Austria
- Universitaire Ziekenhuizen, Leuven, Belgium
- Klinik und Poliklinik für Hautkrankheiten, Sauerbruchstraße, Greifswald, Mecklenburg-Vorpommern, Germany
- Nij Smellinghe Hosptial, Drachten, Netherlands